CLINICAL TRIAL: NCT00609869
Title: A Phase II Study of Lenalidomide (REVLIMID®) in Combination With Rituximab for Patients With CD5+/CD20+ Hematologic Malignancies Who Relapse or Progress After Rituximab
Brief Title: Lenalidomide in Comb w/Rituximab for Pts w/CD5+/CD20+ Hem Malignancies Who Relapse/Progress After Rituximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14978; RV-CLL-PI-067 (Other: Celgene)
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Lymphocytic Leukemia; Mantle Cell Lymphoma
MeSH Terms: conditions — Leukemia, Lymphoid; Lymphoma, Mantle-Cell | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide and Rituximab (Experimental): 28 day cycles of Lenalidomide administered orally and Rituximab administered intravenously.
  Lenalidomide: Escalating doses starting with of 2.5 mg daily on 28-days cycles.
  Rituximab: at 375 mg/m^2 on a weekly basis for the first cycle starting on day 15.
  Interventions: Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide was administered orally with escalating doses on 28-days cycles. The first cycle was administered with a starting dose of 2.5 mg daily on days 1-7, 5mg on days 8-14 and 10 mg on days 15-21, followed by seven days off. On cycle 2 and beyond lenalidomide was administered at 20 mg daily on days 1-21.
  Other Names: REVLIMID®
Drug: Rituximab — Rituximab was administered at 375 mg/m^2 intravenously on a weekly basis for the first cycle starting on day 15. Subsequent rituximab doses were administered on day one of cycle 2 and beyond, every 4 weeks. Doses were repeated on 28-day cycles until disease progression or unacceptable toxicity, but were planned for 12 cycles.
  Other Names: RITUXAN®

SUMMARY:
The purpose of this research is to evaluate the use of Rituximab in combination with Revlimid in the treatment of refractory Mantle Cell Lymphoma (MCL) and Chronic Lymphocytic Leukemia (CLL). Revlimid® is a drug that changes the immune system and it may also get in the way with the growth of tiny blood vessels that help support tumor growth. Therefore, in theory, it may reduce or prevent the growth of cancer cells. Revlimid® is approved by the Food and Drug Administration (FDA) for the treatment of specific types of Myelodysplasia syndrome (MDS) and Multiple Myeloma, two different types of blood cancer. It is currently being tested in a variety of cancer conditions. In this case it is considered experimental.

DETAILED DESCRIPTION:
This phase II trial will use a Simon's two stage design enrolling a total of 28 subjects. Ten will be accrued during stage 1 and 18 during stage 2. If 3 or fewer responses (CR+PR) are observed during the first stage then the trial is stopped early. Given that the 'true' response probability is 30%, there is a 64.96% probability of ending the trial during stage 1. However, if the 'true' response probability is 60% then there is a 5.48% probability that the trial will be stopped in stage 1. If more than 3 responses are observed in stage 1, another 18 patients will be accrued in stage 2. If 12 or fewer responses are observed by the end of the trial, then no further investigation of the drug is warranted. Otherwise, conclude that the drug is worthy of further investigation. The alpha level of the design is 0.04 and the power is 0.91.

Patients with confirmed CD5+/CD20+ MCL or CLL who have relapsed or progressed after Rituximab therapy following a minimum of 6 months duration of response (SD, PR, or CR as defined by Appendix D) will be eligible for this study. Baseline evaluation of patients prior to enrollment in this study will include complete blood counts (CBCs), serum chemistries, liver function tests, kidney function tests, lactate dehydrogenase (LDH); and CT scans of the chest, abdomen and pelvis; and bone marrow biopsy. The exact values for the status of organ function allowable on this protocol are included in the body of this document. Bone marrow aspirates, biopsies and standard FISH evaluation for specific cytogenetic abnormalities will be obtained by the clinical site. An adequate bone marrow aspirate sample is required for a subject to be eligible to participate in this study. All assessments will be completed according to Schedule of Study Assessments.

Patients who meet eligibility criteria and have signed the informed consents will have further laboratory evaluation which will involve flow cytometry of the peripheral blood to evaluate: 1) CD20 density on the leukemic cells (CLL patients only), 2) the percentage of CD56+ cells to evaluate the baseline level of natural killer (NK) cell, 3) the density of activation antigens (CD2, CD11a, CD31, CD38, and CD69) on CD56+ cells, and 4) CD38 (ZAP-70) expression. Pretreatment serum baseline values for Interferon-alpha (IFN-alpha), Tumor necrosis factor-alpha (TNF-A), granulocyte-macrophage colony-stimulating factor (GM-CSF), IL-6, and soluble IL-2 receptor will be obtained. A baseline CBC, flow cytometry and cytokine studies will be obtained on Day 1 prior to start of Lenalidomide.

All patients will have a full immunological evaluation on Day 15 of Lenalidomide therapy prior to Rituximab administration. A bone marrow biopsy will be performed on all patients (CLL and MCL) with prior documented bone marrow involvement once between Days 13- 15 to assess the impact of the lenalidomide on the malignant cells and the surface density of CD20 for patients with CLL before the administration of Rituximab. Flow cytometry on the aspirate specimen will be performed at Moffitt Cancer Center. The cytokine studies will be drawn on Day 15, prior to the administration of Rituximab. Starting on Day 15 after collection of specimens, the patients will receive four weekly doses of Rituximab (375 mg/m^2) concurrent with lenalidomide as per the cycle schedule. Lenalidomide therapy will be continued until progression of disease, unacceptable toxicity or patient withdrawal.

Patient assessment during the clinical trial will be performed by a physician and will occur prior to the administration of each dose of Rituximab. The evaluation will include CBC, routine chemistries, kidney function, liver function, and LDH. The impact of the treatment on any lymphadenopathy or splenomegaly will be documented. Any toxicities noted during these evaluations will be noted. After the four weekly doses of Rituximab, if the pretreatment bone marrow biopsy was positive, the patient will have a repeat bone marrow biopsy to assess response. If the patient had splenomegaly or lymphadenopathy prior to entry into the trial, the patient will need repeat CT scans to assess response. The scans and bone marrow biopsies should be performed two weeks after the patient's last dose of Rituximab.

Follow-up of patients after completing the Rituximab treatment for patients who have not progressed while on therapy will involve a CBC, routine chemistries, liver function tests, and LDH drawn according to the Schedule of Assessments.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed CD5+/CD20+ B-Cell Chronic Lymphocytic Leukemia or Mantle Cell Lymphoma
* Meet the following CLL criteria to participate in this study:

  * Absolute lymphocyte count > 5000/μL
  * CD20+ and CD5+
  * Atypical cells representing < 55% on the peripheral smear
  * Bone marrow lymphocytes ≥ 30%
  * Or previous confirmed diagnosis of CLL/small lymphocytic lymphoma (SLL) with less than 5000/μl or less than 30% lymphocytes in BM
* CLL Patients are eligible if they have stage III or IV disease. Patients with stage 0, I or II disease will be eligible if they have evidence of active disease defined as one or more of the following signs/symptoms:

  * Documented weight loss of ≥ 10% over a six month period
  * Febrile episodes of 38 degrees Celsius (100.5 degrees F) or greater for greater than 2 weeks without evidence of infection
  * Massive or progressive splenomegaly defined as > 6 cm below the left costal margin
  * Massive (> 10 cm in longest diameter) or progressive lymphadenopathy
* Patients with progressive lymphadenopathy will need a biopsy of the lymphadenopathy within the previous six months to ensure that the disease entity remains chronic lymphocytic leukemia. Lymph node biopsy can be deferred if the patient does not have superficial lymphadenopathy that is easily accessible by surgery or by CT guided biopsy.
* The diagnosis of MCL is based upon the National Comprehensive Cancer Network (NCCN) guidelines. The patient's will have biopsy proven CD5+/CD20+/CD23- mantle cell lymphoma with the characteristic cytogenetic abnormality t(11;14) or a cyclin D1 positive immunophenotype. If malignancy is CD23+ but FISH positive for t(11;14), diagnosis of mantle cell lymphoma can be made. Patients with mantle cell lymphoma require appropriate staging which would include upper and lower endoscopy within 2 months of enrollment per NCCN guidelines without additional treatment since the endoscopies.
* Patients with MCL and CLL will be eligible if they have relapsed or progressive disease after Rituximab therapy or a combination therapy including Rituximab. Any other number of previous treatments is allowed including autologous or allogeneic bone marrow transplantation. Patients who are younger than age 65 who have not had a bone marrow transplant must be ineligible or have declined a bone marrow (BM) transplant to participate in this study. Although a transplant is not the standard of care for this patient population, it does provide the best opportunity for a cure.
* Anticipated life expectancy of > 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Baseline organ and marrow function as follows:

  * Absolute neutrophil count ≥1,500/µL
  * Platelets ≥50,000/µL
  * Total bilirubin ≤2.0 mg/dL (34 µmol/L)
  * aspartic transaminase (AST)/alanine transaminase (ALT) ≤2.5 X institutional upper limit of normal(ULN)
  * Creatinine < institutional ULN OR
  * Creatinine clearance ≥60 mL/min/m² for patients with creatinine levels above institutional ULN
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®. Women of childbearing potential, and men with a partner of childbearing potential must follow pregnancy test and birth control guidelines outlined for this study.
* Ability to understand and the willingness to sign a written informed consent document
* Able to adhere to the study visit schedule and other protocol requirements
* Patients with uric acid levels > ULN at baseline must be corrected to ≤ULN prior to the initiation of study therapy.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* May not be receiving any other investigational agents
* Known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lenalidomide and/or thalidomide
* Prior desquamating (blistering) rash with thalidomide
* Neuropathy ≥ grade 2
* Uncontrolled intercurrent illness including (not limited to) ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness/social situations that would limit compliance with study requirements.
* Women currently pregnant or breastfeeding
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* History of another malignancy besides CLL or MCL who have been disease-free ≤ 3 years with exception of basal cell or squamous cell carcinoma of skin or carcinoma in situ of cervix or breast
* Any serious medical condition or psychiatric illness that will prevent patient from signing the informed consent form or will place the patient at unacceptable risk if he/she participates in the study
* Prior use of lenalidomide
* Prior severe hypersensitivity to Rituximab or other murine products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-10; Primary Completion 2014-02 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Pinilla, M.D., PhD., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - Center for Cancer Care & Research/Watson, Lakeland, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Moffitt Cancer Center from October 31, 2007 to March, 22, 2012.
Groups:
- Experimental: Lenalidomide and Rituximab: 28 day cycles of Lenalidomide administered orally and Rituximab administered intravenously.
  Lenalidomide: Escalating doses starting with of 2.5 mg daily on 28-days cycles.
  Rituximab: at 375 mg/m^2 on a weekly basis for the first cycle starting on day 15.
Period: Overall Study
Arm/Group | Experimental: Lenalidomide and Rituximab
Started | 29
Completed | 18
Not Completed | 11
Not completed — Withdrawn, ischemic stroke | 1
Not completed — Severe hematologic toxicity | 1
Not completed — Withdrawal by Subject | 1
Not completed — Seizures | 1
Not completed — Severe tumor flare reaction | 1
Not completed — Hepatitis B infection | 1
Not completed — Rituximab reaction prior to lenalidomide | 1
Not completed — Mantle cell: not evaluable | 4

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Experimental: Lenalidomide and Rituximab
Number analyzed (Participants) | 29
Age, Continuous [Mean (Full Range); unit: years] | 63 [41 to 80]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: The sum of Complete Remission (CR) plus Partial Remission (PR) rates. Duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, and must be confirmed greater than 8 weeks after first meeting CR or PR criteria. Response and progression for Chronic Lymphocytic Leukemia (CLL) were evaluated using 2008 updated National Cancer Institute-Sponsored Working Group Guidelines (NCI-WG) for Chronic Lymphocytic Leukemia. CR: all of the criteria must be met, and patients have the lack disease-related constitutional symptoms: PR: at least two of the criteria of Group A plus one of the criteria of group B have to be met. Group A Parameters: Lymphadenopathy; Hepatomegaly; Splenomegaly; Blood; Lymphocytes; Marrow. Group B Parameters: Platelet count; Hemoglobin; Neutrophils.
Time Frame: Up to 6 years
Population: All evaluable chronic lymphocytic leukemia participants
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Lenalidomide and Rituximab
Number analyzed (Participants) | 18
percentage of participants | 61

2. Secondary Outcome: Clinical Benefit Rate
Description: The ORR rate plus Stable Disease (SD). NCI-WG: SD is the absence of progressive disease (PD) and failure to achieve at least a PR; PD: at least one of the criteria of Group A or Group B has to be met.
Time Frame: Up to 6 years
Population: All evaluable chronic lymphocytic leukemia participants
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Lenalidomide and Rituximab
Number analyzed (Participants) | 18
percentage of participants | 83.3

3. Secondary Outcome: Median Time to Treatment Failure (TTF)
Description: The time from start of therapy to death, Progressive Disease (PD) or initiation of next therapy. PD: at least one of the NCI-WG criteria of Group A or Group B has to be met.
Time Frame: Up to 6 years
Population: All evaluable chronic lymphocytic leukemia participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Lenalidomide and Rituximab
Number analyzed (Participants) | 18
months | 17.7 [5.6 to 29.8]

ADVERSE EVENTS:
Time Frame: 6 years, 3 months
Description: All participants
Arm/Group | Experimental: Lenalidomide and Rituximab
Serious Adverse Events (participants affected / at risk) | 19/29
Other Adverse Events (participants affected / at risk) | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Lenalidomide and Rituximab (N=29)
Hemoglobin - low (Blood and lymphatic system disorders) | 5 (5)
Neutrophils/granulocytes (ANC/AGC) - low (Blood and lymphatic system disorders) | 3 (3)
Platelets - low (Blood and lymphatic system disorders) | 2 (2)
Cardiac Arrhythmia - Other, AFib (Cardiac disorders) | 1 (1)
Cardiac General - Other, AFib/AFlu (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (4)
Fever (in the absence of neutropenia) (General disorders) | 3 (3)
Rigors/chills (General disorders) | 2 (2)
Death not associated with CTCAE term - Death (General disorders) | 1 (1)
Death not associated with CTCAE term - Disease progression NOS (General disorders) | 1 (1)
Dermatology/Skin - Other, dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other, cholilethiasis, gallbladder surgery (Gastrointestinal disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 1 (1)
Infection with Grade 3 or 4 neutrophils - Bladder (urinary) (Infections and infestations) | 1 (1)
Infection with Grade 3 or 4 neutrophils - Blood (Infections and infestations) | 1 (1)
Infection with Grade 3 or 4 neutrophils - Brain + Spinal cord (encephalomyelitis) (Infections and infestations) | 1 (1)
Infection with Grade 3 or 4 neutrophils - Lung (pneumonia) (Infections and infestations) | 6 (9)
Infection with Grade 3 or 4 neutrophils - Upper airway NOS (Infections and infestations) | 1 (1)
Infection - Other, Port A Cath (Infections and infestations) | 5 (7)
Infection - Other, unketiology (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Blood (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 ANC or Grade 1 or 2 (Infections and infestations) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 6 (9)
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (2)
Memory impairment (Nervous system disorders) | 1 (1)
Mental status (Psychiatric disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Pain - Abdomen NOS (General disorders) | 2 (4)
Pain - Chest wall (General disorders) | 1 (1)
Pain - Chest/thorax NOS (General disorders) | 2 (2)
Pain - Neck (General disorders) | 2 (2)
Pain - Pain NOS (General disorders) | 1 (1)
Pain NOS - Back (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal/Genitourinary - Other, chronic renal insufficiency (Renal and urinary disorders) | 1 (1)
Syndromes - Other, tumor fever (General disorders) | 1 (1)
Tumor flare (General disorders) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1)
Vascular - Other, CVA/CNS ischemia (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Lenalidomide and Rituximab (N=29)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 23 (70)
Rigors/chills (General disorders) | 12 (17)
Fever (in the absence of neutropenia) (General disorders) | 11 (14)
Sweating (diaphoresis) (General disorders) | 11 (19)
Insomnia (General disorders) | 7 (11)
Weight loss (General disorders) | 4 (6)
Constitutional Symptoms - (Gastrointestinal disorders) | 18 (36)
Nausea (Gastrointestinal disorders) | 12 (16)
Gastrointestinal - Other (Gastrointestinal disorders) | 10 (13)
Constipation (Gastrointestinal disorders) | 8 (11)
Vomiting (Gastrointestinal disorders) | 7 (9)
Anorexia (Gastrointestinal disorders) | 5 (7)
Distension/bloating, abdominal (Gastrointestinal disorders) | 2 (3)
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 2 (2)
Pain - Other (General disorders) | 14 (43)
Pain - Back (General disorders) | 10 (21)
Pain - Head/headache (General disorders) | 10 (16)
Pain - Abdomen NOS (General disorders) | 6 (11)
Pain - Chest/thorax NOS (General disorders) | 5 (8)
Pain - Lymph node (General disorders) | 5 (8)
Pain - Lymph node (General disorders) | 5 (9)
Pain - Neck (General disorders) | 5 (9)
Pain - Extremity-limb (General disorders) | 4 (8)
Pain - Throat/pharynx/larynx (General disorders) | 4 (4)
Pain - Chest wall (General disorders) | 3 (4)
Pain - Joint (General disorders) | 3 (5)
Pain - Oral cavity (General disorders) | 2 (3)
Pain - Pain NOS (General disorders) | 2 (2)
Pain - Stomach (General disorders) | 2 (2)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 12 (28)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 9 (23)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 4 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (34)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 11 (14)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 8 (21)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) - low (Blood and lymphatic system disorders) | 11 (52)
Hemoglobin low (Blood and lymphatic system disorders) | 8 (13)
Platelets - low (Blood and lymphatic system disorders) | 8 (23)
Lymphopenia (Blood and lymphatic system disorders) | 2 (17)
Infection - Other (Infections and infestations) | 10 (19)
Febrile neutropenia (Infections and infestations) | 8 (10)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 6 (6)
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 4 (6)
Infection with Grade 3 or 4 neutrophils - Lung (pneumonia) (Infections and infestations) | 3 (3)
Infection with unknown ANC - Bronchus (Infections and infestations) | 2 (2)
Infection with unknown ANC - Sinus (Infections and infestations) | 2 (2)
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 2 (2)
Dizziness (Nervous system disorders) | 7 (9)
Neuropathy: sensory (Nervous system disorders) | 7 (14)
Neurology - Other (Nervous system disorders) | 6 (11)
Mood alteration - Anxiety (Psychiatric disorders) | 4 (5)
Mood alteration - Depression (Psychiatric disorders) | 4 (4)
Memory impairment (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 3 (3)
Edema: limb (Blood and lymphatic system disorders) | 13 (21)
Lymphatics - Other (Blood and lymphatic system disorders) | 4 (4)
Edema: head and neck (Blood and lymphatic system disorders) | 2 (6)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 8 (14)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 3 (3)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2 (6)
Vision-blurred vision (Eye disorders) | 5 (6)
Ocular/Visual - Other (Eye disorders) | 4 (5)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Allergic reaction/hypersensitivity (Immune system disorders) | 2 (2)
Hot flashes/flushes (Endocrine disorders) | 4 (6)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 2 (2)
Renal/Genitourinary - Other (Renal and urinary disorders) | 3 (5)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (4)
Hypotension (Cardiac disorders) | 3 (3)
Tumor flare (General disorders) | 3 (4)
Auditory/Ear - Other (Ear and labyrinth disorders) | 3 (6)
Secondary Malignancy - possibly related to cancer treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)

LIMITATIONS AND CAVEATS:
The 4 Mantle Cell participants were not evaluated for Outcome Measures due to their low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes